CLINICAL TRIAL: NCT01541904
Title: STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PRO-118 OPHTHALMIC SOLUTION IN ALLERGIC CONJUNCTIVITIS
Brief Title: Efficacy and Safety of PRO-118 Ophthalmic Solution in Allergic Conjunctivitis
Acronym: PRO-118
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Reformulation
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LVO1209FII; PRO-118
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Ocular Itching; Ocular Allergy; Seasonal Allergic Conjunctivitis; Perennial Allergic Conjunctivitis; Conjunctivitis, Allergic
Keywords: Ocular Allergy.; Seasonal Allergic Conjunctivitis; Perennial Allergic Conjunctivitis; Conjunctivitis, Allergic; Ocular Antihistamines.
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm A. PRO-118/Placebo 0.015%,0.020% (Experimental)
  Interventions: Drug: PRO-118 Ophthalmic Solution 0.015%
- Arm B. PRO-118/Placebo 0.015%,0.020% (Experimental)
  Interventions: Drug: PRO-118 Ophthalmic Solution 0.015 %
- Arm C. PRO-118/Placebo 0.015%,0.020% (Experimental)
  Interventions: Drug: PRO-118 Ophthalmic Solution 0.020 %
- Arm D. PRO-118/Placebo 0.015%,0.020% (Experimental)
  Interventions: Drug: PRO-118 Ophthalmic Solution 0.020 %
- Arm E PRO-118/Placebo 0.015%,0.020% (Placebo Comparator)
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: PRO-118 Ophthalmic Solution 0.015% — PRO-118 Ophthalmic Solution 0.015 % applied qd during 21 days
  Arms: Arm A. PRO-118/Placebo 0.015%,0.020%
Drug: PRO-118 Ophthalmic Solution 0.015 % — PRO-118 Ophthalmic Solution 0.015 % applied twice to day during 21 days
  Arms: Arm B. PRO-118/Placebo 0.015%,0.020%
Drug: PRO-118 Ophthalmic Solution 0.020 % — PRO-118 Ophthalmic Solution 0.020 % applied qd during 21 days
  Arms: Arm C. PRO-118/Placebo 0.015%,0.020%
Drug: PRO-118 Ophthalmic Solution 0.020 % — PRO-118 Ophthalmic Solution 0.020 % applied twice to day during 21 days
  Arms: Arm D. PRO-118/Placebo 0.015%,0.020%
Drug: Placebo Ophthalmic Solution — Placebo Ophthalmic Solution applied qd during 21 days
  Arms: Arm E PRO-118/Placebo 0.015%,0.020%

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of four doses of PRO-118 ophthalmic solution ophthalmic solution compared with placebo, for the treatment of seasonal (SAC) and perennial (PAC) allergic conjunctivitis.

DETAILED DESCRIPTION:
A phase II, double-masked, randomized, placebo-controlled, parallel-group and multicenter clinical trial, to evaluate and compared the clinical efficacy and safety of four doses of PRO-118 ophthalmic solution ( PRO-118 0.015% qd, PRO-118 0.015% twice daily , PRO-118 0.020% qd, PRO-118 0.020% twice daily) for the treatment of seasonal (SAC) and perennial (PAC) allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of seasonal or perennial allergic conjunctivitis.
* Age ≥ 6 years old at screening visit.
* Male or female patients.

Applicable in patients ≥ 18 years old.

* Patient has signed the Informed Consent Form (ICF) prior to any screening procedures.

Applicable in patients with age ≤ 18 years old.

* Patients Patients'parents or legal guardians signed an Informed Consent Form (ICF).
* The patients also provided written assent.

Exclusion Criteria:

* Presence of any form of allergic conjunctivitis other than seasonal or perennial allergic conjunctivitis (Atopic keratoconjunctivitis, giant papillary conjunctivitis).
* Any other ophthalmic medication within seven days prior to randomization.
* Patient with one blind eye.
* Visual acuity of 20/40 in any eye.
* Patients with history of active stage of any other concomitant ocular disease.
* Contraindications or sensitivity to any component of the study treatments.
* Contact lens users.
* Ocular surgery within the past 3 months.
* Women who were not using an effective means of contraception or who were pregnant or nursing.
* Participation in any studies of investigational drugs within 90 days previous to the inclusion.

Discontinuation criteria:

* Patients could be discontinued before the completion of the study because of use of prohibited medications, adverse events, pregnancy, protocol violations, lack of efficacy, or administrative reasons.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of PRO-118 ophthalmic solution. | 21 days.
  Primary efficacy measure: Evaluation of ocular itching.
  Secondary efficacy measures: Evaluation of symptoms(redness eye,ocular irritation, foreign body sensation, photophobia and lacrimation) and signs(conjunctival hyperaemia,chemosis, mucous discharge ocular and presence of follicles/papillae).

SECONDARY OUTCOMES:
Safety of PRO-118 Ophthalmic Solution. | 21 days.
  * Evaluation of ocular symptoms and signs, visual acuity (VA), biomicroscopy, intraocular pressure (IOP), funduscopy and cup disc-ratio.
  * Frequency, severity and relationship to study medication of all adverse events occurring during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: María C Jiménez-Martínez, MD, Principal Investigator — "Instituto de Oftalmología Fundación Conde de Valenciana, I.A.P."; Concepción Santacruz-Valdés, MD, Principal Investigator — "Instituto de Oftalmología Fundación Conde de Valenciana, I.A.P."; Emma T Villaseñor-Fierro, MD, Principal Investigator — Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde"; Miriam Becerra-Cotta, MD, Principal Investigator — Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde"; Leopoldo M Baiza-Durán, MD, Study Director — Clinical Research Department. Laboratorios Sophia SA de CV
Locations (2):
- Mexico (2):
  - Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - "Instituto de Oftalmología Fundación Conde de Valenciana, I.A.P, Mexico City